CLINICAL TRIAL: NCT06524778
Title: The Therapeutic Effect of Single High-dose Brachytherapy for Locally Inoperable and Metastatic Giant Osteosarcoma Masses
Brief Title: Single High-dose Brachytherapy for Giant Osteosarcoma Masses
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Jiao Tong University Affiliated Sixth People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaojing Yang, Principal Investigator, Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSH06R102
Record Dates: First submitted 2024-07-24; First posted 2024-07-29 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Osteosarcoma
Keywords: brachytherapy; high-dose; osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Brachytherapy

STUDY DESIGN:
Intervention Model Description: Single dose high-dose （10Gy）implantable brachytherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- brachytherapy (Experimental): Patients with locally unresectable giant osteosarcoma masses who meet the criteria are enrolled in the experimental group, and all patients receive a single dose of 10Gy of implantable brachytherapy. Record treatment-related acute events during and after treatment. Follow up on survival and local control after treatment ends, marking the end of the trial treatment.
  Interventions: Radiation: brachytherapy

INTERVENTIONS:
Radiation: brachytherapy — Patients with locally unresectable giant osteosarcoma masses who meet the criteria are enrolled in the experimental group, and all patients receive a single dose of 10Gy of implantable brachytherapy. Record treatment-related acute events during and after treatment. Follow up on survival and local control after treatment ends, marking the end of the trial treatment.

SUMMARY:
This study is a prospective, single-arm, phase II, single-center study. Patients with locally unresectable giant osteosarcoma masses who meet the criteria are enrolled in the experimental group, and all patients receive a single dose of 10Gy of implantable brachytherapy. Record treatment-related acute events during and after treatment. Follow up on survival and local control after treatment ends, marking the end of the trial treatment.

DETAILED DESCRIPTION:
Screening period: Local MRI or CT examination, blood routine and coagulation function test.

Selected treatment period: All enrolled patients received one dose of close range interstitial radiotherapy with a radiation dose of 10 Gy. The number of insertion needles depends on the size and location of the tumor. The instrument used for radiotherapy is the Medda high-dose rate brachytherapy machine, and the radiation source is 192 iridium. Record treatment related acute events such as bleeding during the treatment period.

Follow up: Follow up with local MRI or CT at 1 month, 3 months, 6 months, and 1 year after the end of radiotherapy treatment to evaluate the treatment effect; Simultaneously follow up with patients for survival and treatment related adverse reactions, such as dermatitis, infections, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosis of osteosarcoma;
2. Age range 12-70 years old;
3. The primary or metastatic lesion cannot be surgically removed based on clinical evaluation, and treatment with internal medicine multi line chemotherapy, targeted therapy, immunotherapy, etc. is ineffective;
4. ECOG physical fitness status is 0-1 points;
5. According to RECIST version 1.1 standard, there must be at least one evaluable target lesion with a mass length diameter greater than 5cm;
6. Sign a written informed consent form before conducting any experimental activities;
7. Researchers determine that they are able to comply with the research protocol;
8. Patients who are willing and able to comply with visit arrangements, treatment plans, laboratory tests, and other research procedures.

Exclusion Criteria:

1. Local mass previously received radiation therapy;
2. Major surgery ≤ 4 weeks before enrollment;
3. Previous or concurrent malignant tumors (excluding malignant tumors that have been cured and have a cancer free survival of more than 5 years, such as basal cell carcinoma of the skin and papillary thyroid carcinoma);
4. Pregnant or lactating women;
5. Active pulmonary tuberculosis.

Ages: 12 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 6 months
  6 months of progression-free survival

SECONDARY OUTCOMES:
progression-free survival | 12 months
  12 months progression-free survival
progression-free survival | 12 months
  12 months of progression-free survival
OS | 12 months
  12 months of OS
Adverse reactions related to radiotherapy | 12 months
  Adverse reactions

IPD SHARING:
Plan to Share IPD: Undecided
No.